CLINICAL TRIAL: NCT04385732
Title: Melanoma Surveillance Photography (MSP) to Improve Early Detection of Melanoma in Ultra-high and High Risk Patients
Acronym: IMAGE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Melanoma and Skin Cancer Trials Limited (Other)
Collaborators: Monash University (Other); University of Sydney (Other); The University of Queensland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 02.19
Record Dates: First submitted 2020-04-01; First posted 2020-05-13 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2024-11

CONDITIONS: Melanoma; Skin Cancer; Anxiety and Fear
Keywords: Dermatology; Teledermatology; 2D Total Body Imaging; 3D Total Body Imaging; Melanoma Surveillance Photography; Biopsy; Excision; Health-related Quality of Life; Health system utilisation; Health economics
MeSH Terms: conditions — Melanoma; Skin Neoplasms; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The trial is an open-label, multi-site, parallel-arm randomised controlled trial. Participants meeting the eligibility criteria will be randomised 1:1 to either standard care or the intervention arm. Randomisation will be 1:1 to either Intervention or Control group stratified by high/ultra-high risk of 2nd primary melanoma, sex, 2D/3D imaging, GP/Dermatologist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care plus Melanoma Surveillance Photography (Experimental): Clinical surveillance standard of care with addition of 2D or 3D Melanoma Surveillance Photography and digital dermoscopy.
  Interventions: Device: 2D or 3D Melanoma Surveillance Photography
- Standard of Care (No Intervention): Clinical surveillance standard of care without Melanoma Surveillance Photography.

INTERVENTIONS:
Device: 2D or 3D Melanoma Surveillance Photography — Total body imaging using 2D or 3D Melanoma Surveillance Photography plus digital dermoscopy.
  Arms: Standard of Care plus Melanoma Surveillance Photography

SUMMARY:
This randomised controlled trial will investigate the role of melanoma surveillance photography (MSP) in the surveillance of patients at high or ultra-high risk of melanoma. MSP is a comprehensive method of melanoma monitoring which includes total body photography and digital dermoscopy which is performed at prescribed intervals. The study will test whether participants under surveillance with MSP have less unnecessary biopsies (false positives) compared to those without MSP. Participants will be Australian residents with a new diagnosis of primary melanoma, who have multiple naevi and are at high or ultra-high risk of developing melanoma. Participants will be randomised 1:1 to either groups.

It is hypothesised that those randomised to surveillance with MSP will have better patient outcomes. Improved diagnostic performance as measured by the number of unnecessary biopsies will be the primary outcome measure.

DETAILED DESCRIPTION:
The primary aim is to test whether melanoma surveillance with MSP, comprising either 2D or 3D TBP tagged with digital dermoscopy, compared to clinical surveillance without MSP, results in improved diagnostic performance, specifically reduced number of unnecessary biopsies (i.e. false positives due to an excision or biopsy of a lesion being performed to diagnose melanoma and that lesion being identified on pathology as benign), in high (and very high) risk individuals whose risk is contributed to by high naevus counts.

The secondary aims are to:

1. Evaluate whether MSP:

   1. Results in improved sensitivity of doctors' diagnosis of melanoma (i.e. reduction in false negatives)
   2. Improves health-related quality of life, patient satisfaction, and reduces patient anxiety
   3. Reduces costs to patients and health care system
2. Evaluate the safety and acceptability of MSP
3. Evaluate benefit of MSP in high risk patients prior to a primary melanoma diagnosis (Sub-study 1)
4. Evaluate diagnostic performance of tele-dermatology compared to en-face clinical visits (Sub-study 2).

Investigators hypothesise that for ultra-high and high risk patients with multiple naevi, clinical surveillance with melanoma surveillance photography (compared to without MSP) will lead to better patient outcomes, in particular a reduction in the number of unnecessary biopsies (i.e. false positives) as a measure of diagnostic performance. Secondary hypotheses include that for ultra-high, and high risk patients with multiple naevi, clinical surveillance with MSP (compared to without MSP) will lead to:

1. Reduction in the number of misclassified melanoma malignancies (i.e. false negatives);
2. Reduction in the number of misclassified melanocytic and keratinocyte lesions combined;
3. Improved quality of life; and
4. Favourable health economic outcomes.

ELIGIBILITY:
Inclusion criteria

Patients may be included in the study if they meet ALL of the following criteria:

1. Aged 18 years or older at date of diagnosis
2. Within 24 months (2 years) of the date of diagnosis when attending Screening & Baseline Visit: where date of diagnosis refers to the date on the pathology report that provides histological confirmation of primary cutaneous melanoma (insitu or invasive)
3. Able to provide informed consent, complete questionnaires, and attend trial site for MSP*
4. Appropriate for TBP referral
5. High/very high risk of subsequent primary melanoma (see risk assessment tool, Appendix IV)*
6. Multiple naevi, as "some" or "many" naevi on pictogram below at Screening & Baseline visit.
7. Not previously under active surveillance (at least yearly) with TBP for melanoma surveillance (see inclusion criteria 9)
8. Living in Australia and not planning to move overseas within the next 3 years
9. Participants that meet all eligibility criteria but have previously been under active surveillance with TBP for at least the previous 2 years meet exclusion critierion 1, in which case they are ineligible for the main study and eligible for sub-study 1 only.

   Active surveillance with TBP refers to TBP images having been taken AND used for melanoma surveillance. As such, if a patient had TBP but these images were not used for melanoma surveillance (i.e. not used by clinicians to monitor a patient's skin), then surveillance is not considered active and the patient would still be eligible for the main study (as well as sub-study 1).
10. Patients need to have had at least annual surveillance over the past 2 years (at least) to be eligible for sub-study 1 (note that this refers to annual skin surveillance not annual TBP images being taken) (i.e. do not meet inclusion criteria 7 are eligible for sub-study 1)

Exclusion criteria

Patients will be excluded from the study for ANY of the following reasons:

1. Previously under active surveillance with TBP (active surveillance referring to TBP images being used for melanoma surveillance Stage IV metastatic melanoma
2. Stage IV metastatic melanoma
3. Ocular melanoma, mucosal melanoma
4. Participation in another clinical trial or study involving MSP

Note:

A past history of other cancers is not an exclusion criteria.

*These eligibility criteria cannot be assessed by the cancer registry. These criteria will be assessed by the study team and/or referring doctor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 670 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of melanoma surveillance | 24 months
  The primary outcome is the diagnostic performance of surveillance for melanoma, expressed as the number of false positive biopsies per patient over a 24-month period.

SECONDARY OUTCOMES:
Cost-effectiveness of MSP | 24 months
  Standard health economic cost-effectiveness measures.
Diagnostic performance for melanoma | 24 months
  Agreement and reliability indices.
Diagnostic performance for keratinocyte lesions | 24 months
  Agreement and reliability indices.
Health-Related Quality of life | 24 months
  Assessment of Quality of Life (AQOL-8D) questionnaire for calculation of quality-adjusted life years (QALYs). Minimum score per each of 8 questions is 1; maximum score is 5, where higher score represents worse outcomes. Scores may be aggregated to provide an overall index of the health state utility per participant, where higher scores indicate worse quality of life outcomes.
Patient anxiety | 24 months
  European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30), Fear of Cancer Recurrence - short form (FCR4) and a purpose-designed patient acceptability scale will be utilised to synthesise a single endpoint measure for patient anxiety. Value range is 0 to 100, where higher values represent greater anxiety (worse outcomes).

OTHER OUTCOMES:
IMAGE Sub-study 1: PRE-TRIAL EXCISION RATES | 5 year (retrospective)
  To estimate the benefit of MSP in high risk patients prior to a melanoma diagnosis, amongst participants who would have been classified as 'high risk' at the time of their primary melanoma, this sub-study will compare:
  i) Breslow thickness of the primary melanoma at entry into this trial, and ii) Biopsy rates prior to diagnosis
IMAGE Sub-study 2: TELEDIAGNOSIS VALIDATION | Validity analysis undertaken at a single time point based on data accrued over 24 month study period.
  Approximately 100 paired sets of 3D surveillance and digital dermoscopy images (baseline and follow-up) taken from patients in the intervention arm, will be sent to 10 participating study doctors (both GPs and dermatologists; all 100 pairs sent to all 10 doctors) for teledermatology assessment. The study doctors will assess the images with respect to whether they have a melonama present or not. Images will be selected randomly from amongst patients accrued to the main study for this telediagnosis validation study. Approximately 30% of these will include an image of a melanoma confirmed by histopathology (gold standard) during the trial. This substudy will not affect patient care but will assess diagnostic performance (sensitivity and specificity) in the teledermatology setting compared to the en-face clinical setting in order to validate the use of telediagnosis in routine care.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Mar, Principal Investigator — Monash University and Alfred Health
Locations (12):
- Australia (12):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Newcastle Skin Check, Newcastle, New South Wales
  - Dermatology Clinical Trials Unit, Westmead Hospital, Sydney, New South Wales
  - Melanoma Institute Australia, Wollstonecraft, New South Wales
  - Diamantina Institute, University of Queensland, Brisbane, Queensland
  - FNQH Cairns Skin Cancer Centre, Cairns, Queensland
  - Skin Repair Skin Cancer Clinic, Townsville, Townsville, Queensland
  - Bendigo Cancer Centre Research Unit, Bendigo Health, Bendigo, Victoria
  - Skin Health Institute, Carlton, Victoria
  - Phillip Island Health Hub, Bass Coast Health, Cowes, Victoria
  - Victorian Melanoma Service, Alfred Health, Melbourne, Victoria
  - Wonthaggi Hospital, Bass Coast Health, Wonthaggi, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yan MK, Cust AE, Soyer HP, Janda M, Loewe K, Byars G, Fishburn P, White P, Mahumud RA, Saw RPM, Herschtal A, Fernandez-Penas P, Guitera P, Morton RL, Kelly J, Wolfe R, Mar VJ. Study protocol for a randomised controlled trial to evaluate the use of melanoma surveillance photography to the Improve early detection of MelanomA in ultra-hiGh and high-risk patiEnts (the IMAGE trial). Trials. 2023 Mar 29;24(1):236. doi: 10.1186/s13063-023-07203-5. PMID 36991460
- See also: Detailed information on the IMAGE trial — https://www.masc.org.au/image/